CLINICAL TRIAL: NCT06716671
Title: Influence of Continuous Glucose Monitoring on Quality of Life in People With Type 2 Diabetes Mellitus
Acronym: Glucocavi
Status: Active, not recruiting | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Sergi Rodríguez Soler, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: 24/166-P
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Continuous Glucose Monitoring; Quality of Life; Type 2 Diabetes Mellitus (T2DM)
Keywords: Continuous Glucose Monitoring; Quality of Life; Primary Care; Hypoglycemia; Type 2 Diabetes Mellitus; Patient satisfaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Type 2 diabetes and continuous glucose monitoring Tarragona: People with type 2 diabetes and intensive insulin therapy who are using a continuous glucose monitoring sensor for the first time in the Camp de Tarragona health region.

SUMMARY:
Background: Diabetes Mellitus (DM) is a chronic disease that affects millions of people worldwide. More than 95% of cases are type 2 diabetes mellitus (T2DM). In recent years, diabetes management has evolved with the introduction of continuous glucose monitoring (CGM) devices. These devices implanted under the skin allow continuous measurement of glucose levels monitoring glucose trends and the rate at which glucose level rise and fall without the need for capillary glycaemias test. While studies demostrate the effectiveness of CGM devices in controlling glucose levels in adults with T2DM, there is no evidence related to quality of life in this patients.

Hypothesis: The use of CGM in people with T2DM improves their quality of life, reduces distress about the disease, reduces fear of hypoglycaemia, increases detection of hypoglycaemia, and improves metabolic control.

Objectives: To assess quality of life, diabetes distress, fear of hypoglycaemia, detection of hypoglycaemia, and metabolic control in people with T2DM before and after the use of CGM sensors.

Methodology: Prospective observational pre-post unblinded study. Adults with type 2 diabetes using a CGM device in the primary care setting will be followed for 12 months. They will be asked to complete 5 questionnaires at baseline, and 4 questionnaires at 3, 6 and 12 months. No other activity that differs from usual clinical practice will be performed.

Data analysis: a descriptive analysis of the main study variables will be carried out and the differences in the data before and after the intervention will be analysed using the chi-square test for qualitative variables, and the Student's t-test for quantitative variables. Statistical significance will be accepted at a p-value < 0.05.

Applicability and relevance: The results of the study will provide information on whether CGM devices improve quality of life and glycaemic control in people with type 2 diabetes. With these results it will be possible to assess whether it is beneficial to extend funding for CGM devices to more of the population than is currently the case.

DETAILED DESCRIPTION:
Study development: The recruitment period runs from September 2024 to February 2025. Participants will be recruited by health professionals (nurse or doctor) CGM referents from each of the 20 primary care centres in the Camp de Tarragona health region. Sampling will be by convenience, all persons who meet the inclusion criteria and none of the exclusion criteria will be offered to participate in the study. Participants must sign an informed consent and their data will be coded.

Participants will be asked to fill in 5 questionnaires at the beginning of the study:

* Sociodemographic questionnaire created ad hoc to know the profile of the patients.
* EsDQOL questionnaire that assesses the quality of life related to diabetes.
* DDS17 questionnaire that assesses diabetes-related distress.
* EsHFS questionnaire that assesses fear of hypoglycaemia.
* Clarke Test that assesses the detection of hypoglycaemia.

The EsDQOL, DDS17, EsHFS and Clarke Test questionnaires must be repeated at 3, 6 and 12 months after the start of the study. Participants will be called to their primary care centre of reference to fill in the questionnaires themselves and these will be kept on paper at the centre until data analysis.

To assess metabolic control, the data provided by the CGM sensor will be used and the results of the AGP (Ambulatory Glucose Profile) report of the first 2 weeks will be compared with the data at 3, 6 and 12 months. No analytical tests or capillary blood glucose measurements will be requested.

Data analysis: A descriptive analysis of the main study variables will be performed using percentages for qualitative variables and mean and standard deviation for quantitative variables. To analyse the differences in the data before and after the intervention, chi-square tests will be used for qualitative variables and the Student's t-test for quantitative variables. Statistical significance will be accepted with a p-value <0.05. Data will be analysed using SPSS statistical software version 23 or later.

Sample calculation: Accepting an alpha risk of 0.05 and a statistical power greater than 0.8 in a bilateral contrast, 55 subjects are required to detect as statistically significant a difference equal to or greater than 9 units in the EsDQOL questionnaire (main study variable). A common standard deviation of 23.65 is estimated. A loss to follow-up rate of 0% is estimated. [GRANMO sample size calculator v7.10 available at Calculator (laalamedilla.org)].

ELIGIBILITY:
Inclusion Criteria:

* Treatment with intensive insulin therapy (basal bolus regimen with 3 or more daily doses of insulin).
* Perform 6 or more daily capillary glycaemia determinations.
* Be willing to use a CGM device for at least 70% of the time.
* Undergo training on the use of the CGM device by the centre's CGM referent.
* Agree to participate in the study.

Exclusion Criteria:

* Cognitive impairment measured by Pfeiffer test with a score of 3 or more errors.
* Previous use of a CGM device.
* Pregnancy.
* Being institutionalised.
* Having participated in another research study related to diabetes mellitus within the last year.
* Not having proper handling of the CGM device: inability to download glycaemic control data, inability to keep the sensor attached to the skin, not understanding how it works, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is adults in an industrialised country with a diagnosis of type 2 diabetes with intensive insulin regimen who will start using a CGM sensor. Participants will be recruited from primary care centres in the Camp de Tarragona health region following inclusion and exclusion criteria. Depending on the location of the primary care centre, the population may be from an urban, semi-urban, or rural setting.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference between pre and post "diabetes-related quality of life (EsDQOL)" questionnaire. | 0, 3, 6 and 12 months
  A validated scale is used to measure diabetes-related quality of life. It consists of 43 questions with answers on a Likert scale from 1 to 5. The higher the score, the worse the quality of life.

SECONDARY OUTCOMES:
Difference between pre and post "diabetes-related distress scale (DDS17)". | 0, 3, 6 and 12 months
  A validated scale is used to measure diabetes-related distress. It consists of 17 questions with answers on a Likert scale from 1 to 6. An average score < 2 points is considered normal, moderate distress a score between 2.0 and 2.9 points, and high distress a score equal to or higher than 3.
Difference between pre and post "hypoglycaemia fear test (EsHFS)". | 0, 3, 6 and 12 months
  A validated scale is used to measure the hypoglycaemia fear. It consists of 24 questions with answers on a Likert scale from 1 to 5. The higher the score, the greater the fear of hypoglycaemia.
Difference between pre and post "undetected hypoglycemia test (Test de Clarke)". | 0, 3, 6 and 12 months
  A validated test that assesses the patient's ability to detect hypoglycaemia. Each response is classified as normal or abnormal. If the sum total of abnormal responses is ≥4, the patient has an abnormal perception of hypoglycaemia, 3 abnormal responses is considered undetermined, and 2 or less is considered normal perception.
Difference between pre and post metabolic control. | 2 weeks, 3 months, 6 months, 12 months.
  The CGM sensor provides several metabolic control values: % time glucose in range (70-180mg/dl), % time between 70mg/dl and 54mg/dl, % time below 54mg/dl, % time between 180mg/dl and 250mg/dl, % time above 250mg/dl, average glucose, glucose management indicator (GMI), and glucose variability (%CV). Data from the patient's first AGP report 2 weeks after starting to use the CGM sensor will be compared with data at 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Rodríguez-Soler, Nurse, Principal Investigator — Institut Català de la Salut
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Chesser H, Srinivasan S, Puckett C, Gitelman SE, Wong JC. Real-Time Continuous Glucose Monitoring in Adolescents and Young Adults With Type 2 Diabetes Can Improve Quality of Life. J Diabetes Sci Technol. 2024 Jul;18(4):911-919. doi: 10.1177/19322968221139873. Epub 2022 Nov 23. PMID 36416098
- [Background] Moreno-Fernandez J, Gomez FJ, Galvez Moreno MA, Castano JP. Clinical Efficacy of Two Different Methods to Initiate Sensor-Augmented Insulin Pumps: A Randomized Controlled Trial. J Diabetes Res. 2016;2016:4171789. doi: 10.1155/2016/4171789. Epub 2016 Nov 29. PMID 28004007
- [Background] Gilbert TR, Noar A, Blalock O, Polonsky WH. Change in Hemoglobin A1c and Quality of Life with Real-Time Continuous Glucose Monitoring Use by People with Insulin-Treated Diabetes in the Landmark Study. Diabetes Technol Ther. 2021 Mar;23(S1):S35-S39. doi: 10.1089/dia.2020.0666. PMID 33470882
- [Background] Gehlaut RR, Dogbey GY, Schwartz FL, Marling CR, Shubrook JH. Hypoglycemia in Type 2 Diabetes--More Common Than You Think: A Continuous Glucose Monitoring Study. J Diabetes Sci Technol. 2015 Apr 27;9(5):999-1005. doi: 10.1177/1932296815581052. PMID 25917335
- [Background] Rodriguez de Vera Gomez P, Mateo Rodriguez C, Rodriguez Jimenez B, Hidalgo Sotelo L, Peinado Ruiz M, Torrecillas Del Castillo E, Ruiz-Aranda D, Serrano Olmedo I, Candau Martin A, Martinez-Brocca MA. Impact of Flash Glucose Monitoring on the Fear of Hypoglycemia Phenomenon in Adults with Type 1 Diabetes. Diabetes Technol Ther. 2024 Jul;26(7):478-487. doi: 10.1089/dia.2023.0370. Epub 2024 Feb 22. PMID 38315507
- [Background] Charleer S, Mathieu C, Nobels F, De Block C, Radermecker RP, Hermans MP, Taes Y, Vercammen C, T'Sjoen G, Crenier L, Fieuws S, Keymeulen B, Gillard P; RESCUE Trial Investigators. Effect of Continuous Glucose Monitoring on Glycemic Control, Acute Admissions, and Quality of Life: A Real-World Study. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1224-1232. doi: 10.1210/jc.2017-02498. PMID 29342264
- [Background] Rodbard D. Continuous Glucose Monitoring: A Review of Recent Studies Demonstrating Improved Glycemic Outcomes. Diabetes Technol Ther. 2017 Jun;19(S3):S25-S37. doi: 10.1089/dia.2017.0035. PMID 28585879
- [Background] Kieu A, King J, Govender RD, Ostlundh L. The Benefits of Utilizing Continuous Glucose Monitoring of Diabetes Mellitus in Primary Care: A Systematic Review. J Diabetes Sci Technol. 2023 May;17(3):762-774. doi: 10.1177/19322968211070855. Epub 2022 Feb 1. PMID 35100891
- [Background] Hirsch IB. Introduction: History of Glucose Monitoring. In: Role of Continuous Glucose Monitoring in Diabetes Treatment. Arlington (VA): American Diabetes Association; 2018 Aug. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK538968/ PMID 34251770
- [Background] McGill JB, Ahmann A. Continuous Glucose Monitoring with Multiple Daily Insulin Treatment: Outcome Studies. Diabetes Technol Ther. 2017 Jun;19(S3):S3-S12. doi: 10.1089/dia.2017.0090. PMID 28585875